CLINICAL TRIAL: NCT01112397
Title: A Phase I, Open-Label, Multi-Center, Dose-Escalation Study to Assess the Safety and Tolerability, and Pharmacokinetics of AZD1480 Administered as Daily Oral Monotherapy in Patients With Advanced Solid Malignancies in the Escalation Phase and EGFR or ROS Mutant NSCLC or Non-Smokers With Lung Metastasis in the Expansion Phase.
Brief Title: Study to Assess Safety, Tolerability and PK of AZD1480 in Patients With Solid Tumours
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Decision to stop development of AZD1480
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D1060C00002
Record Dates: First submitted 2010-04-23; First posted 2010-04-28 (Estimated); Last update posted 2013-07-22 (Estimated); Status verified 2013-07

CONDITIONS: Solid Malignancies
Keywords: Jak2; cancer; jak 1; stat 3; Phase 1
MeSH Terms: conditions — Neoplasms | interventions — AZD 1480

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): AZD1480 until Maximum Tolerated Dose (MTD) is reached
  Interventions: Drug: AZD1480
- 2 (Experimental): AZD1480 dose expansion of MTD
  Interventions: Drug: AZD1480

INTERVENTIONS:
Drug: AZD1480 — continuous daily oral capsule

SUMMARY:
This study is being conducted to assess the safety, tolerability and PK of AZD1480 in patients with advanced solid malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced solid cancer without available therapy in the escalation phase and mutation positive NSCLC or non-smokers with other primary tumors lung metastasis in the expansion phase
* ECOG Performance Status 0-1
* Evidence of post-menopausal status in females or males willing to use barrier contraception

Exclusion Criteria:

* Prior therapy with any JAK2 medications
* Significant lung disorder or lung disease. Previous radiation therapy to chest wall or chest infection requiring antibiotic treatment within 21 days before study screening. Evidence of significant pulmonary hypertension or COPD
* Eye disease of the cornea

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2010-04; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability as assessed by Adverse events, vital signs, ECGs, Pulmonary Function Tests (DLco, FEV, FVC, Oxygen saturation) and laboratory data (chemistry, hematology and Urinalysis) | Information will be collected from the time the informed consent is signed, throughout the study

SECONDARY OUTCOMES:
Evaluation of the pharmacokinetics of AZD1480 | During all cycles

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Curt, MD, Study Chair — AstraZeneca
Locations (3):
- United States (3):
  - Research Site, Aurora, Colorado
  - Research Site, Detroit, Michigan
  - Research Site, Philadelphia, Pennsylvania